CLINICAL TRIAL: NCT04344535
Title: Convalescent Plasma to Reduce Complications Associated With COVID-19 Infection: A Randomized Trial Comparing the Efficacy and Safety of High-Titer Anti-SARS-CoV-2 Plasma vs. Standard Plasma in Hospitalized Patients With COVID- 19 Infection
Brief Title: Convalescent Plasma vs. Standard Plasma for COVID-19
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Insufficient eligible and consenting patients
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Elliott Bennett-Guerrero, Professor of Anesthesiology, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SBU-COVID19-ConvalescentPlasma
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Results first posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: COVID

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Staff in Transfusion Services (Blood Bank) at Stony Brook will be unblinded so they can collect, store, and dispense either convalescent plasma or standard plasma. They will affix an approved label with all required information, e.g. bar code, blood type, expiration date, and will indicate that the bag contains convalescent plasma/standard plasma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Convalescent Donor Plasma (Active Comparator)
  Interventions: Biological: Convalescent Plasma
- Standard Donor Plasma (Placebo Comparator)
  Interventions: Biological: Standard Donor Plasma

INTERVENTIONS:
Biological: Convalescent Plasma — 450-550 mL of plasma containing anti-SARS-CoV-2 antibody titer ideally > 1:320, but meeting minimum titer per FDA Guidelines for convalescent plasma.
  Arms: Convalescent Donor Plasma
Biological: Standard Donor Plasma — 450-550 mL of plasma with low titer to anti-SARS-CoV-2 antibodies
  Arms: Standard Donor Plasma

SUMMARY:
The purpose of this study is to find out if transfusion of blood plasma containing antibodies against COVID-19 (anti-SARS-CoV-2), which were donated from a patient who recovered from COVID-19 infection, is safe and can treat COVID-19 in hospitalized patients.

Antibodies are blood proteins produced by the body in response to a virus and can remain in the person's bloodstream (plasma) for a long time after they recover. Transferring plasma from a person who recovered from COVID-19 may help neutralize the virus in sick patients' blood, and/or reduce the chances of the infection getting worse.

ELIGIBILITY:
There are 2 groups of research subjects: plasma donor and recipients

Volunteer plasma donors can donate Convalescent Plasma if they:

* have adequate antibody levels against COVID-19 per FDA Guidelines
* have had no symptoms of COVID-19 for at least 14 days
* meet routine plasma donation criteria

Inclusion Criteria for Plasma Recipients:

* Adults 18 years of age or older
* Hospitalized with PCR+ COVID-19 infection
* If female must not be pregnant and/or breastfeeding.

Exclusion Criteria for Plasma Recipients:

* Unable to randomize patient within 14 days of admission to Stony Brook Hospital (or any other hospital if a transfer to Stony Brook Hospital).
* In the treating physician's opinion, the patient cannot tolerate a 450-550 mL infusion of plasma over up to 8 hours (4 hours max per unit), even if prophylaxed with intravenous diuretic
* Contraindication to transfusion or history of prior reactions to blood transfusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Bennett-Guerrero, MD, Principal Investigator — Stony Brook Hospital
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub6. PMID 37162745
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 Feb 1;2(2):CD013600. doi: 10.1002/14651858.CD013600.pub5. PMID 36734509
- [Derived] Piechotta V, Iannizzi C, Chai KL, Valk SJ, Kimber C, Dorando E, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 May 20;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub4. PMID 34013969
- [Derived] Bennett-Guerrero E, Romeiser JL, Talbot LR, Ahmed T, Mamone LJ, Singh SM, Hearing JC, Salman H, Holiprosad DD, Freedenberg AT, Carter JA, Browne NJ, Cosgrove ME, Shevik ME, Generale LM, Andrew MA, Nachman S, Fries BC; Stony Brook Medicine COVID Plasma Trial Group; Stony Brook Medicine COVID Plasma Trial Group are as follows: Investigators; Principal Investigator, Critical Care; Pathology/Blood Bank; Infectious Disease; Safety Monitor; Biostatistics; Hematology; (Blood Bank; and; Pathology, Laboratory Services). Team 1 (Online Survey/In Person Scheduling); Team Leader; and; Team 2 (In Person Screening Visits); Team Leader; and; Team 3 (Patient/Recipient Screening, Plasma Administration, Data Capture); Team Leader; and; and; and; and; Team M (Antibody Testing/Randomization):; Team Leader; and; Plaque Reduction Neutralization Assay: Janet Hearing. Regulatory (Investigational New Drug [IND] and Institutional Review Board [IRB] support); (IND support); (IRB support), and; Data and Safety Monitoring Board (DSMB); and; (Chair) and; (unblinded DSMB statistician); Stony Brook Medicine COVID Plasma Trial Group and Stony Brook Medicine COVID Plasma Trial Group are as follows: Investigators and Principal Investigator, Critical Care and Pathology/Blood Bank and Infectious Disease and Safety Monitor and Biostatistics and Hematology and (Blood Bank and and and Pathology, Laboratory Services). Team 1 (Online Survey/In Person Scheduling) and Team Leader and and and Team 2 (In Person Screening Visits) and Team Leader and and and Team 3 (Patient/Recipient Screening, Plasma Administration, Data Capture) and Team Leader and and and and and and and and and Team M (Antibody Testing/Randomization): and Team Leader and and and Plaque Reduction Neutralization Assay: Janet Hearing. Regulatory (Investigational New Drug [IND] and Institutional Review Board [IRB] support) and (IND support) and (IRB support), and and Data and Safety Monitoring Board (DSMB) and and and (Chair) and and (unblinded DSMB statistician). Severe Acute Respiratory Syndrome Coronavirus 2 Convalescent Plasma Versus Standard Plasma in Coronavirus Disease 2019 Infected Hospitalized Patients in New York: A Double-Blind Randomized Trial. Crit Care Med. 2021 Jul 1;49(7):1015-1025. doi: 10.1097/CCM.0000000000005066. PMID 33870923

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 8 screen failures prior to randomization, thus 74 patients were randomized.
Period: Overall Study
Arm/Group | Convalescent Donor Plasma | Standard Donor Plasma
Started | 59 | 15
Completed | 59 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Convalescent Donor Plasma | Standard Donor Plasma | Total
Number analyzed (Participants) | 59 | 15 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] — years
  years | 67 (15.8) | 64 (17.4) | 66 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 7 | 30
  Male | 36 | 8 | 44
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 42 | 8 | 50
  Black | 5 | 1 | 6
  Other | 12 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: 28 Day Ventilator Free Days
Description: Number of days a patient is receiving mechanical invasive ventilation through 28 days post randomization. Patients who die during this time period are assigned 0 ventilator free days.
Time Frame: 28 days post randomization
Population: All randomized
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Convalescent Donor Plasma | Standard Donor Plasma
Number analyzed (Participants) | 59 | 15
days | 28 [2 to 28] | 28 [0 to 28]

2. Secondary Outcome: 90 Day All-cause Mortality
Description: All cause mortality from randomization until 90 days post randomization
Time Frame: 90 days
Population: All randomized
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Donor Plasma | Standard Donor Plasma
Number analyzed (Participants) | 59 | 15
Participants | 16 | 5

ADVERSE EVENTS:
Time Frame: Adverse Events (death, infusion reaction requiring termination of study plasma infusion, or Grade 4 or greater Organ Failure) were collected for the first 28 days. All-cause mortality was also assessed at 90 days.
Description: Adverse Events (death, infusion reaction requiring termination of study plasma infusion, or Grade 4 or greater Organ Failure) were collected for the first 28 days. All-cause mortality was also assessed at 90 days.
Arm/Group | Convalescent Donor Plasma | Standard Donor Plasma
All-Cause Mortality (participants affected / at risk) | 16/59 | 5/15
Serious Adverse Events (participants affected / at risk) | 8/59 | 1/15
Other Adverse Events (participants affected / at risk) | 0/59 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Convalescent Donor Plasma (N=59) | Standard Donor Plasma (N=15)
Renal Failure (Renal and urinary disorders) | 5 | 0 — Grade 4 or greater Renal Failure
Pulmonary Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 — Grade 4 or greater Pulmonary Failure
Liver Failure (Hepatobiliary disorders) | 3 | 0 — Grade 4 or greater Liver Failure
Hematologic Failure (Blood and lymphatic system disorders) | 1 | 1 — Grade 4 or greater Hematologic Failure
Infusion Reaction (Blood and lymphatic system disorders) | 1 | 0 — Infusion reaction resulting in termination of study plasma infusion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-16): https://cdn.clinicaltrials.gov/large-docs/35/NCT04344535/Prot_SAP_000.pdf